CLINICAL TRIAL: NCT03096769
Title: Ergonomics in Robotic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John A. Occhino, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-009275
Record Dates: First submitted 2017-03-21; First posted 2017-03-30 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Musculoskeletal Strain; Ergonomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Other)
  Interventions: Other: Ergonomist

INTERVENTIONS:
Other: Ergonomist — The intervention consists of each surgeon meeting with an ergonomist where the ergonomist will adjust the console settings and chair height to an ergonomically optimal position.

SUMMARY:
This study is designed to answer if an ergonomist can configure a daVinci robot console to improve surgeon discomfort. Adjustments to the robot console will be surgeon specific as they are tailored to their individual body type. Measurements will be taken at the time of console configuration.

ELIGIBILITY:
Inclusion Criteria:

* Fellowship trained, specialty board certified gynecologic surgeon.
* Robot used for hysterectomy until completion of vaginal cuff closure.

Exclusion Criteria:

- Any non-robotic method to perform hysterectomy (laparotomy, non-robotic laparoscopic, vaginal approach).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Nordic Upper Body Questionnaire Score | Baseline, Immediately postoperative (approximately one hour)
  The Nordic upper body questionnaire will be one measure of upper body musculoskeletal discomfort following robotic hysterectomy.
Change in Body Part Discomfort Questionnaire Score | Baseline, Immediately postoperative (approximately one hour)
  The Body Part Discomfort Questionnaire will be one measure of upper body musculoskeletal discomfort following robotic hysterectomy
Surgical Task Load Index Score | Immediately postoperative (approximately one hour)
  The surgical task load index score will be one measure of upper body musculoskeletal discomfort following robotic hysterectomy.

SECONDARY OUTCOMES:
Change in measurement of console settings (in cm) | Baseline, up to 1 year
  Comparison between surgeon- and ergonomist-derived console settings
Change in measurement of console head angle (in degrees) | Baseline, up to 1 year
  Comparison between surgeon- and ergonomist-derived console settings

CONTACTS AND LOCATIONS:
Overall Officials: John A Occhino, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No